CLINICAL TRIAL: NCT00395902
Title: A Retrospective Evaluation of Sensipar Use in Renal Transplant Recipients
Brief Title: Post Transplant Study
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Other Study IDs: 20040261; 2004261
Record Dates: First submitted 2006-11-02; First posted 2006-11-06 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Kidney Tansplant; Secondary Hyperparathyroidism; Hyperparathyroidism
Keywords: Sensipar; cinacalcet; Mimpara
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Hyperparathyroidism

STUDY DESIGN:
Time Perspective: Retrospective

INTERVENTIONS:
Drug: Sensipar after Post Transplant

SUMMARY:
Retrospective chart review to gather information on Sensipar patterns of use and effects on biochemical parameters in renal transplant recipients

ELIGIBILITY:
Inclusion Criteria:

* Adults >= 18 years old
* Subjects who have received Sensipar for a duration of at least 3 months, beginning at least 3 months after a kidney transplant. Subjects must have begun Sensipar teatment no later than Februry 28, 2005 at treating physician's discretion.

Exclusion Criteria:

* Subjects who received Sensipar before undergoing a kidney transplant
* Subjects receiving dialysis post-transplant

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com